CLINICAL TRIAL: NCT07394699
Title: Efficiency of Intermittent Hypoxia Intervention in Primary Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IH-PI
Record Dates: First submitted 2024-05-05; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Insomnia, Primary
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IH group (Active Comparator): Participants will receive 10 times intermittent hypoxia (oxygen concentration: 13%) intervention.
  Interventions: Other: Intermittent Hypoxia
- Control group (Sham Comparator): Participants will receive 10 times sham-hypoxia (oxygen concentration: 21%) intervention in 5 days.
  Interventions: Other: Sham Intermittent Hypoxia

INTERVENTIONS:
Other: Intermittent Hypoxia — The intermittent hypoxia protocol refers to four cycles of 5 minutes hypoxia inhaling interval by 5 minutes normoxia, which is performed twice a day (at least 6 hours apart) in 7 days.
  Arms: IH group
Other: Sham Intermittent Hypoxia — The sham intermittent hypoxia protocol refers to 45 minutes normoxia inhaling, which is performed twice a day (at least 6 hours apart) in 7 days.
  Arms: Control group

SUMMARY:
The purpose of this study was to understand the effectiveness of intermittent hypoxia in the treatment of primary insomnia.

DETAILED DESCRIPTION:
Insomnia is a sleep disorder characterized by frequent and persistent difficulties in falling asleep or maintaining sleep, and resulting in inadequate sleep satisfaction. Insomnia is a common sleep problem with a prevalence of 10% to 15% in adults and a chronic course that may increase with age, with nearly half of those with severe insomnia lasting more than 10 years.Insomnia can increase the risk of some diseases, such as anxiety, depression, hypertension, diabetes and cardiovascular diseases. Insomnia is closely related to the body's chronic inflammatory response, and studies have shown that insomnia induces a chronic inflammatory response in the body, which impairs the structure and integrity of sleep, leading to an increased inflammatory response in the body, which in turn impairs the health.

Intermittent hypoxia (IH) refers to periodic hypoxic-normoxic training performed with brief exposure to hypoxia. Previous studies have shown that short-term intermittent hypoxia can produce neuroprotective effects, inhibit inflammatory response, and promote neurological recovery, providing a new approach for the treatment of primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are diagnosed with primary insomnia between 18 and 60 years old，gender is not limited.
* Patients who are not taking sedative-hypnotic drugs or have stopped taking drugs for more than 2 weeks.
* Residing in the plains all year round and not having been above 1500 meters above sea level in the past 30 days.
* Quiet state SaO2 ≥ 90%, cerebral oxygen saturation 58-82%, heart rate 60-100 beats/min, blood pressure 90-140/60-90 mmHg, respiratory rate 16-20 times/min.
* No functional drinks, caffeine-containing beverages, or sleep-disturbing medications during the study period.

Exclusion Criteria:

* Stroke onset in the past 3 months, other severe neurological diseases, such as epilepsy, intracranial infectious diseases or demyelination.
* Uncontrolled hypertension (systolic blood pressure ≥200mmHg) with antihypertensive drugs before enrollment, other cardiovascular diseases.
* History of pulmonary, hepatic, dermatologic, or hematologic diseases.
* History of substance abuse.
* Pregnancy, Severe sleep apnea and neurological disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The polysomnography between IH group and control group | Baseline and Day 7
  Before and after the experiment, polysomnography was performed on both the experimental and control groups to record sleep latency, total sleep duration, as well as the duration and proportion of each sleep stage.

SECONDARY OUTCOMES:
Concentration of serum parameters between IH group and control group | Baseline and Day 7
  Measure tumor markers, IL-6, IL-1β, and other relevant indicators in both the experimental and control groups before and after the experiment.
The score of Insomnia Severity Index（ISI） | Baseline and Day 7
  The Insomnia Severity Index (ISI) total score is included as a separate secondary outcome measure, with values on a scale ranging from 0 to 28, where higher scores indicate a worse outcome (greater severity of insomnia).
The score of the Flinders Fatigue Scale (FFS) | Baseline and Day 7
  The Flinders Fatigue Scale (FFS) total score is included as a separate secondary outcome measure, with values on a scale ranging from 0 to 31, where higher scores indicate a worse outcome (greater fatigue severity).
The scale of Self-Rating Anxiety Scale (SAS) | Baseline and Day 7
  The Self-Rating Anxiety Scale (SAS) total score is included as a separate secondary outcome measure, with values on a scale ranging from 25 to 100, where higher scores indicate a worse outcome (higher levels of anxiety).
The score of Self-Rating Depression Scale (SDS) | Baseline and Day 7
  The Self-Rating Depression Scale (SDS) total score is included as a separate secondary outcome measure, with values on a scale ranging from 25 to 100, where higher scores indicate a worse outcome (higher levels of depression).
Peripheral Oxygen Saturation (SpO₂) | Day 1-7
  The Peripheral Oxygen Saturation (SpO₂) is included as a separate outcome measure, with values on a percentage scale ranging from 0% to 100%, where higher scores indicate a better outcome (higher level of blood oxygenation).
Heart Rate | Day 1-7
  The Heart Rate is included as a separate outcome measure, measured in beats per minute (bpm). While there is no universal fixed range, values are assessed against normal clinical reference ranges, where extreme values (either too high or too low) indicate a worse outcome.
Respiratory Rate | Day 1-7
  The Respiratory Rate is included as a separate outcome measure, measured in breaths per minute (brpm). While there is no universal fixed range, values are assessed against normal clinical reference ranges, where extreme values (either too high or too low) indicate a worse outcome.
Blood Pressure | Day 1-7
  Blood Pressure is included as a separate outcome measure, measured in millimeters of mercury (mmHg) and reported as the combination of systolic and diastolic values. While there is no universal fixed range, values are assessed against normal clinical reference ranges, where extreme values (either too high or too low) indicate a worse outcome.